CLINICAL TRIAL: NCT02730624
Title: Population Pharmacokinetics and Pharmacodynamics Study of Piperacillin/Tazobactam During Early Phase in Critically Ill Patients With Severe Sepsis
Brief Title: Piperacillin/Tazobactam in Critically Ill Patients With Severe Sepsis and Septic Shock
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sutep Jaruratanasirikul (Other)
Collaborators: Prince of Songkla University (Other)
Responsible Party: Sponsor-Investigator, Sutep Jaruratanasirikul, Principal Investigator, Prince of Songkla University
Organization: Prince of Songkla University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIP-56501141
Record Dates: First submitted 2016-02-24; First posted 2016-04-06 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2016-03

CONDITIONS: Early Phase of Severe Sepsis and Septic Shock
Keywords: piperacillin/tazobactam; critically ill; severe sepsis; septic shock
MeSH Terms: conditions — Shock, Septic; Critical Illness; Sepsis | interventions — Piperacillin, Tazobactam Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- piperacillin/tazobactam (Experimental): 4.5 g of piperacillin/tazobactam in 100 ml of normal saline solution was administered via an infusion pump at a constant flow rate 30 min every 6 h
  Interventions: Drug: Piperacillin-tazobactam

INTERVENTIONS:
Drug: Piperacillin-tazobactam — 4.5 g of piperacillin/tazobactam in 100 ml of normal saline solution was administered via an infusion pump at a constant flow rate 30 min every 6 h and blood sample were obtained by direct venepuncture at 0, 0-0.5, 0.5-2, 2-4 and 4-6 hour after drug administration

SUMMARY:
This is prospective study to assess the pharmacodynamics (t>MIC) of 4.5 g every 6 h of piperacillin/tazobactam in patients with early phase of severe sepsis/septic shock following administration by a 30 min infusion.

Clinical and laboratory data such as age, sex, body weight, electrolyte, vital signs, APACHAE II score, BUN, Cr and fluid balance will be collected.

Fifty patients will be enrolled in this study. Piperacillin pharmacokinetic study will be carried out during the piperacillin/tazobactam therapy.

Each patient received 4.5 g every 6 h of piperacillin/tazobactam within 24 h of severe sepsis or septic shock, blood samples (approximately 3 ml) will be obtained by direct venipuncture at the following time: 0, 0-0.5, 0.5-2, 2-4 and 4-6 h after piperacillin/tazobactam therapy.

Concentration of piperacillin in plasma will be simulated in Monte Carlo technique to get PK/PD index and reported to % PTA and % CFR.

ELIGIBILITY:
Inclusion Criteria:

* sepsis patient (defined by 2011 SCCM/ESICM/ACCP/ATS/SIS International sepsis definition conference)
* severe sepsis or septic sock was defined by

  * Severe sepsis (sepsis with organ dysfunction)
  * Septic shock (sepsis with systolic arterial pressure<90 mmHg, mean arterial pressure<60 mmHg or decrease systolic blood pressure> 40 mmHg from base line)

Exclusion Criteria:

* Patients who are pregnant.
* Patients who have documented hypersensitivity to beta-lactam
* Patients who are dialysis
* Patients who are severe sepsis or septic shock more than 24 hour

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-03; Primary Completion 2016-05 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Concentration of piperacillin in plasma | 6 hour after the piperacillin dose
  Concentration of piperacillin in plasma will be simulated in Monte Carlo simulation to assess PK/PD index as 40% and 100% T>MIC and will be reported as %PTA.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Clinical Pharmacology, Department of Medicine, Faculty of Medicine, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand